CLINICAL TRIAL: NCT03571334
Title: Botulinum Toxin A for the Treatment of Chemotherapy Induced Peripheral Neuropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Erin McGonigle, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ebeddows
Record Dates: First submitted 2018-06-11; First posted 2018-06-27 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy
MeSH Terms: interventions — incobotulinumtoxinA; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IncobotulinumtoxinA (Experimental): IncobotulinumtoxinA (Xeomin®, Merz) (INA) will be reconstituted with preservative-free normal saline to a dilution of 5mL:100 units.
  Study participants in this arm will receive 50u INA (total volume 2.5mL) injected into each limb, max 2 limbs per subject (either bilateral hands or bilateral feet.)
  Hands: INA will be injected across the palmar surface of the digits in a grid like pattern covering a total of 25 sites per limb (0.1mL/site).
  Feet: INA will be injected across the dorsal surface of the feet also in a grid like pattern covering a total of 25 sites per limb (0.1mL/site).
  Interventions: Drug: IncobotulinumtoxinA (Xeomin®, Merz) (INA)
- saline control (Placebo Comparator): Study participants in this arm will 2.5mL normal saline injected into each limb, max 2 limbs per subject (either bilateral hands or bilateral feet.)
  Hands: saline will be injected across the palmar surface of the digits in a grid like pattern covering a total of 25 sites per limb (0.1mL/site).
  Feet: Saline will be injected across the dorsal surface of the feet also in a grid like pattern covering a total of 25 sites per limb (0.1mL/site).
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: IncobotulinumtoxinA (Xeomin®, Merz) (INA) — IncobotulinumtoxinA (Xeomin®, Merz) (INA) will be reconstituted with preservative-free normal saline to a dilution of 5mL:100 units. Study participants will receive 50u INA (total volume 2.5mL) injected into each limb, max 2 limbs per subject (either bilateral hands or bilateral feet.) Study participants will receive one series of injections during the trial. In the hands, INA will be injected across the palmar surface of the digits in a grid like pattern covering a total of 25 sites per limb (0.1mL/site). In the feet, INA will be injected across the dorsal surface of the foot in a grid like pattern covering a total of 25 sites per limb (0.1mL/site). Injections will be performed intradermally using a 5/16-inch, 32-g needle
  Other Names: Xeomin® (Brand name)
  Arms: IncobotulinumtoxinA
Drug: Normal saline — Study participants will total volume 2.5mL of 0.9% Normal saline injected into each limb, max 2 limbs per subject (either bilateral hands or bilateral feet.) Study participants will receive one series of injections during the trial. In the hands, 0.9% Normal saline will be injected across the palmar surface of the digits in a grid like pattern covering a total of 25 sites per limb (0.1mL/site). In the feet, 0.9% Normal saline will be injected across the dorsal surface of the foot in a grid like pattern covering a total of 25 sites per limb (0.1mL/site). Injections will be performed intradermally using a 5/16-inch, 32-g needle
  Arms: saline control

SUMMARY:
Chemotherapy induced peripheral neuropathy (CIPN) is a common side effect of taxanes and platinum derivative based chemotherapeutic agents, common in breast cancer treatment regimens. It can have a significant effect on both quality of life and treatment outcomes, often resulting in dose modifications and early treatment discontinuation. The use of IncobotulinumtoxinA (INA) ((Xeomin®, Merz) has recently been shown to be effective in the treatment of neuropathic pain via inhibiting the release of several neurotransmitters involved in pain signaling pathway.

The purpose of this study is to examine the efficacy and safety of intradermal INA injections for treatment of CIPN in breast cancer patients. The study will recruit a total of 40 participants, randomly assigned to receive either INA (Experimental group, n=20) or saline placebo injections (Control group n=20).

Potential participants who have received chemotherapy for breast cancer will be screened for the diagnosis of peripheral neuropathy. After obtaining informed consent, participants will be further screened with the DN4 questionnaire, a clinician administered questionnaire that has a high level of sensitivity and specificity in discriminating neuropathic pain. Those study participants who score ≥4 on this tool will undergo nerve conduction studies to confirm the presence of peripheral neuropathy. Recruited study participants will then be randomized to treatment or control groups; the treatment group will undergo intradermal injections of INA (100 Units INA, total volume 5ml), and the control groups will undergo placebo injection with preservative-free normal saline (equal volume, 5mL). Total injection volume will be divided evenly and injected intradermally into a total of 50 sites on either the feet or hands (25 sites per limb).

The primary outcome will be the assessment of pain using the neuropathic pain scale (NPS) prior to intervention and at eight weeks post intervention. Secondary outcomes will include the change in NPS for each domain at additional time points: 2weeks, 4 weeks, 12 weeks, 6 months, the change in the Neuropathic Pain Impact on Quality of Life (NePIQoL) score at time points: 2 weeks, 4 weeks, 8 weeks, 12 weeks, 6 months, and the incidence of treatment related adverse events within each cohort. Statistical analysis will be utilized to determine whether the injection of intradermal INA is effective in improving pain as measured by the NPS scales vs placebo.

We hypothesize that the study participants treated with INA will have lower NPS scores as compared to placebo.

DETAILED DESCRIPTION:
Chemotherapy Induced Peripheral Neuropathy Chemotherapy induced peripheral neuropathy (CIPN) is a common adverse effect of cancer therapy, effecting over half of all patients who receive chemotherapy. CIPN typically manifests as a symmetrical, predominately sensory peripheral neuropathy, and is most common in taxanes, vinca-alkaloids, and/or platinum compounds. Taxanes are microtubule stabilizing agents and are effective in the treatment of many solid organ cancers, often used as first line therapy in the treatment of breast cancer. Taxanes cause peripheral neuropathy by injuring neurons, disrupting axonal transport, and causing wide spread macrophage activation both in the periphery as well as at the dorsal root ganglion (DRG) and microglial activation in the spinal cord. The incidence of CIPN is high following taxane administration, and often occurs before patients have completed the prescribed course. In severe cases it can lead to dose modifications and early treatment discontinuation, effecting overall survivorship. Additionally, it has been demonstrated to have a profound effect on quality of life, found to correlate with increased fatigue, malaise, increased psychological distress and a less sense of well being and satisfaction with life. Current treatment options are inadequate, with suboptimal treatment effect size and dose limiting adverse effects. Various neuroprotective regimens have been trialed, including co-administration of thiols, neurotrophic factors, antioxidants and vitamin E; however none of these approaches are consistently effective in reducing peripheral neuropathy.

Botulinum Toxin (BoNT) Botulinum toxin (BoNT) is routinely used to treat a wide variety of disorders, traditionally by decreasing muscle activity through inhibiting the release of acetylcholine from the presynaptic nerve terminal. There has been a recent increase and growing body of evidence for the use of botulinum toxin in the treatment of neuropathic pain including postherpetic neuralgia, diabetic neuropathy, complex regional pain syndrome, trigeminal neuralgia, phantom limb pain, spinal cord injury-induced neuropathic pain, and central post-stroke pain.

The mechanism by which BoNT effects neuropathic pain is independent than the effect of BoNT on muscle relaxation. There are several proposed mechanisms by which BoNT decreases neuropathic pain, all of which likely contributing to the antinociceptive effect. First, it has been shown that BoNT inhibits the release of sensory neurotransmitters such as substance P, calcitonin gene related peptide, and glutamate from nerve endings into the peripheral nerve terminal. This not only directly mediates pain, but has also been shown to result in decreased inflammation. In addition, recent work in the rat model suggests that the antinociceptive mechanism of BoNT may in part be due to a reduction of TRPV1 expression. TRPV1 is a well-known pain receptor which responds to mechanical, thermal and chemical stimuli, is heavily expressed on the DRG. BoNT has been shown to exhibit retrograde axonal transport from the periphery, so effects on the DRG and central nervous system cannot be overlooked and likely play a role in the mechanism.

Recently, intradermal BoNT injections were found efficacious in treating diabetic peripheral neuropathy. Multiple studies have demonstrated a reduction in Visual Analog Scale (VAS) scores following intradermal BoNT injections on the dorsal aspect of the foot in diabetic patients with peripheral neuropathy. Similar to CIPN, diabetic neuropathy presents in a stocking-glove distribution with a predominant sensory neuropathy. BoNT has additionally been proven to be safe and efficacious when used specifically in a cohort of head, neck, and breast cancer patients who developed post surgical and post radiation neuropathic pain. In this study, affected patients underwent intradermal BoNT injections which resulted in improvement in VAS and clinical global impressions of change (CGI-C) scales. Together, this evidence suggests that intradermal BoNT injections are efficacious in the treatment of neuropathic pain, and is safe for use in the cancer population. If our hypothesis proves correct, we will demonstrate the efficacy of BoNT for treatment of CIPN, allowing for improved treatment options. An antihyperalgesic effect following intradermal BoNT injections was additionally observed in rats with Paclitaxel induced peripheral neuropathy, again suggesting that BoNT will be an effective treatment specifically in the CIPN patient population.

In controlled studies, BoNT has consistently demonstrated a minimal adverse effect profile. Typically, adverse effects occur within one week of BoNT injection and are transient. As with any injection, localized pain, infection, bleeding may be associated. A metaanalysis of two studies using BoNT for the treatment of diabetic neuropathic pain concluded that there were no statistically significant adverse effects associated with BoNT treatment. Intradermal injections for the treatment of hyperhidrosis have FDA approval, and the most common adverse events associated (3-10% of adult patients) were injection site pain and hemorrhage.

The specific aim of this study is to determine the efficacy of intradermal INA injections to reduce chemotherapy induced peripheral neuropathy in breast cancer patients who have undergone taxane-based chemotherapy. We hypothesize the treatment group who receives intradermal INA injections will have lower neuropathic pain scale (NPS) scores when compared to the control group who receives saline injections.

1.0 Objective

The purpose of this study is to examine the change in pain via the neuropathic pain scale (NPS) in patients with chemotherapy induced peripheral neuropathy (CIPN) following intradermal IncobotulinumtoxinA ((Xeomin®, Merz) (INA) injections.

2.0 Experimental Design

The study is a prospective, randomized, double-blinded placebo-controlled study. Forty study participants will be enrolled in this study and randomized into Control vs. Experimental groups

1. Study participants will be screened in the breast cancer clinics of Drs. Chitambar and Kamaraju and other breast oncology providers at the Medical College of Wisconsin/Froedtert Hospital for symptoms of Grade II neuropathic pain (per Common Terminology Criteria for Adverse Events [CTCAE] v5.0) thought secondary to chemotherapy.
2. Study participants interested in pursuing the study will be contacted by phone by a study team member and the protocols and consent form will be discussed. Interested participants will be scheduled for an appointment in the translational research unit (TRU) at the Medical College of Wisconsin.

   a. The adult TRU is located within Froedtert Hospital and is dedicated strictly to conducting human research. Facilities include basic medical equipment, fully staffed nursing support, 5 exam rooms and 3 procedure rooms.
3. The study participant will have the opportunity to ask the investigator about any questions they may have. Following this, the consent form will be signed and a copy will be given to the patient.
4. Study participants will then be issued the DN4 questionnaire, a clinician administered questionnaire that has a high level of sensitivity and specificity in discriminating neuropathic pain. A score ≥4 represents likely neuropathic pain.
5. Study participants will then undergo nerve conduction velocity (NCV) exams to confirm diagnosis of sensory neuropathy. Exam will be administered by PM&R physician or resident.
6. Study participants will complete baseline neuropathic pain scale (NPS) assessments
7. Study participants will complete baseline Neuropathic Pain Impact on Quality of Life (NePIQoL) assessment
8. Study participants will disclose and document current pain medication regimen. This will include scheduled and prn medications taken for treatment of chemotherapy induced peripheral neuropathy as well as scheduled and prn medications used for treatment of other nociceptive pain.
9. Recruited participants will then be randomized to Experimental vs Control groups
10. Study participants who meet inclusion criteria will then undergo intradermal injection of INA or placebo into the bilateral hands or feet, depending on the location of the neuropathic pain. The injecting physician, Dr. Erin McGonigle (PI)/Dr. Erin Beddows (Co-I) and the subject will be blinded to the contents of the injection.

    1. INA will be reconstituted with preservative-free normal saline to a dilution of 5mL:100 units
    2. Anatomical site of injections (hands vs feet) will be determined based on patient report of severity of pain and impact of pain on quality of life.
    3. 2% lidocaine jelly will be applied as a topical anesthetic for 3 minutes to site of injections
    4. Site of injections will then be thoroughly cleaned with antiseptic solution of 75% alcohol and allowed to dry

       * Study participants undergoing intradermal injections of bilateral hands/feet will receive 50u INA (total volume 2.5mL) or equivalent volume normal saline injected into each limb, max 2 limbs per subject.
       * INA or saline equivalent will be injected across the palmar surface of the digits in a grid like pattern covering a total of 25 sites per limb (0.1mL/site).
       * INA will be injected across the dorsal surface of the feet also in a grid like pattern covering a total of 25 sites per limb (0.1mL/site).
       * Injections will be performed intradermally using a 5/16-inch, 32-g needle

2.1 Study Duration

* The duration of this study will be 6 months following intervention. 2.2 Study Participants Responsibilities
* Study participants will need to attend one research-related clinic visit for NCS testing
* Study participants will need to attend one research-related clinic visit for injection

  o This may be the same visit as the NCS
* Study participants will be requested to answer a telephone and/or RedCap survey pending the participant's preference.

2.3 Study participants

* Forty study participants will be enrolled in this double blinded, randomized, controlled trial and they will be grouped by treatment method: Experimental vs. Control, as determined by a randomization table
* Study participants will be over 18 years of age, both genders, all ethnicities, and currently diagnosed with chemotherapy induced peripheral neuropathy

ELIGIBILITY:
Inclusion Criteria:

1. Been diagnosed with breast cancer and undergone treatment with taxane based chemotherapeutic agents. Patients with metastatic and non metastatic disease are eligible.
2. Have neuropathic pain with onset within 6 months of chemotherapy
3. Must score >4 on DN4 scale, a scale with high specificity and sensitivity for differentiating neuropathic pain from somatic and nociceptive pain
4. Age >18 years, male and/or female
5. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. End Stage Renal Disease patients on Hemodialysis
2. Female participants who are pregnant (positive urine pregnancy test), who have an infant they are breastfeeding, or intend to become pregnant within 6 months.
3. History of peripheral neuropathy attributed to any cause other than chemotherapy
4. Currently receiving chemotherapy, or having had received chemotherapy in the past 6 months
5. Prior treatment with Botulinum Toxin A for any indication within the past 6 months
6. Changes in neuropathic pain modulators within 1 month prior to enrollment or during the course of the trial. Participants who require rescue medications for breakthrough pain can be given so at the discretion of their provider.
7. Hypersensitivity reaction to INA injection
8. Distal muscle weakness and/or atrophy
9. Active infection at injection site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in pain from baseline at eight weeks as measured by the change in Neuropathic Pain Scale (NPS) | baseline and 8 weeks
  The primary outcome of this study will be the change pain as measured by the NPS at 8 weeks post intervention as compared to baseline NPS scores. The NPS is a validated scale that is used to classify patient's neuropathic pain. It includes assessment of global pain intensity and pain unpleasantness, two items addressing the location of the pain as deep or surface, and six items addressing the specific qualities of neuropathic such as sharp, hot, dull, cold, sensitivity, and itchy.

SECONDARY OUTCOMES:
Improvement in pain from baseline as measured by the change in Neuropathic Pain Scale (NPS) | baseline and 2 weeks, 4 weeks, 12 weeks, 6 months
  Change pain as measured by the NPS at additional time points: 2weeks, 4 weeks, 12 weeks, 6 months when compared to baseline scores.
Change in pain characteristics as measured by the change in each individual domain of Neuropathic Pain Scale (NPS) | baseline and 2 weeks, 4 weeks, 8 weeks, 12 weeks, 6 months
  Change in the pain characteristics as measured by each NPS domain when compared to baseline at additional time points: 2weeks, 4 weeks, 8 weeks, 12 weeks, 6 months. Domains include: assessment of global pain intensity and pain unpleasantness, two items addressing the location of the pain as deep or surface, and six items addressing the specific qualities of neuropathic such as sharp, hot, dull, cold, sensitivity, and itchy.
Change in quality of life as measured by the Neuropathic Pain Impact on Quality of Life (NePIQoL) score | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 6 months post intervention
  Change in the Neuropathic Pain Impact on Quality of Life (NePIQoL) score at time points: 2 weeks, 4 weeks, 8 weeks, 12 weeks, 6 months. The NePIQoL is a validated scale comprised of 42 items organized into 7 categories of questions affecting quality of life: symptoms, relationships, psychological, social activity, physical change, personal care, overall health and overall quality of life
Safety as measured by self reporting of incidence of treatment related adverse events | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 6 months post intervention
  incidence of treatment related adverse events within each cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apfel SC. Botulinum toxin for neuropathic pain? Neurology. 2009 Apr 28;72(17):1456-7. doi: 10.1212/WNL.0b013e3181a412b2. Epub 2009 Mar 25. No abstract available. PMID 19321845
- [Background] Argyriou AA, Bruna J, Marmiroli P, Cavaletti G. Chemotherapy-induced peripheral neurotoxicity (CIPN): an update. Crit Rev Oncol Hematol. 2012 Apr;82(1):51-77. doi: 10.1016/j.critrevonc.2011.04.012. Epub 2011 Sep 10. PMID 21908200
- [Background] Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, Cunin G, Fermanian J, Ginies P, Grun-Overdyking A, Jafari-Schluep H, Lanteri-Minet M, Laurent B, Mick G, Serrie A, Valade D, Vicaut E. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005 Mar;114(1-2):29-36. doi: 10.1016/j.pain.2004.12.010. Epub 2005 Jan 26. PMID 15733628
- [Background] Cui M, Khanijou S, Rubino J, Aoki KR. Subcutaneous administration of botulinum toxin A reduces formalin-induced pain. Pain. 2004 Jan;107(1-2):125-33. doi: 10.1016/j.pain.2003.10.008. PMID 14715398
- [Background] Fan C, Chu X, Wang L, Shi H, Li T. Botulinum toxin type A reduces TRPV1 expression in the dorsal root ganglion in rats with adjuvant-arthritis pain. Toxicon. 2017 Jul;133:116-122. doi: 10.1016/j.toxicon.2017.05.001. Epub 2017 May 3. PMID 28478059
- [Background] Favre-Guilmard C, Auguet M, Chabrier PE. Different antinociceptive effects of botulinum toxin type A in inflammatory and peripheral polyneuropathic rat models. Eur J Pharmacol. 2009 Sep 1;617(1-3):48-53. doi: 10.1016/j.ejphar.2009.06.047. Epub 2009 Jul 1. PMID 19576881
- [Background] Francisco GE, Tan H, Green M. Do botulinum toxins have a role in the management of neuropathic pain?: a focused review. Am J Phys Med Rehabil. 2012 Oct;91(10):899-909. doi: 10.1097/PHM.0b013e31825a134b. PMID 22660369
- [Background] Freeman R, Wallace MS, Sweeney M, Backonja MM. Relationships Among Pain Quality, Pain Impact, and Overall Improvement in Patients with Postherpetic Neuralgia Treated with Gastroretentive Gabapentin. Pain Med. 2015 Oct;16(10):2000-11. doi: 10.1111/pme.12791. Epub 2015 Jun 25. PMID 26115203
- [Background] Galer BS, Jensen MP. Development and preliminary validation of a pain measure specific to neuropathic pain: the Neuropathic Pain Scale. Neurology. 1997 Feb;48(2):332-8. doi: 10.1212/wnl.48.2.332. PMID 9040716
- [Background] Park HJ, Lee Y, Lee J, Park C, Moon DE. The effects of botulinum toxin A on mechanical and cold allodynia in a rat model of neuropathic pain. Can J Anaesth. 2006 May;53(5):470-7. doi: 10.1007/BF03022619. PMID 16636031
- [Background] Jensen MP, Friedman M, Bonzo D, Richards P. The validity of the neuropathic pain scale for assessing diabetic neuropathic pain in a clinical trial. Clin J Pain. 2006 Jan;22(1):97-103. doi: 10.1097/01.ajp.0000173018.64741.62. PMID 16340598
- [Background] Kottschade LA, Sloan JA, Mazurczak MA, Johnson DB, Murphy BP, Rowland KM, Smith DA, Berg AR, Stella PJ, Loprinzi CL. The use of vitamin E for the prevention of chemotherapy-induced peripheral neuropathy: results of a randomized phase III clinical trial. Support Care Cancer. 2011 Nov;19(11):1769-77. doi: 10.1007/s00520-010-1018-3. Epub 2010 Oct 9. PMID 20936417
- [Background] Lakhan SE, Velasco DN, Tepper D. Botulinum Toxin-A for Painful Diabetic Neuropathy: A Meta-Analysis. Pain Med. 2015 Sep;16(9):1773-80. doi: 10.1111/pme.12728. Epub 2015 Mar 20. PMID 25800040
- [Background] Lucioni A, Bales GT, Lotan TL, McGehee DS, Cook SP, Rapp DE. Botulinum toxin type A inhibits sensory neuropeptide release in rat bladder models of acute injury and chronic inflammation. BJU Int. 2008 Feb;101(3):366-70. doi: 10.1111/j.1464-410X.2007.07312.x. PMID 18184328
- [Background] Mols F, Beijers T, Vreugdenhil G, van de Poll-Franse L. Chemotherapy-induced peripheral neuropathy and its association with quality of life: a systematic review. Support Care Cancer. 2014 Aug;22(8):2261-9. doi: 10.1007/s00520-014-2255-7. Epub 2014 May 1. PMID 24789421
- [Background] Park J, Park HJ. Botulinum Toxin for the Treatment of Neuropathic Pain. Toxins (Basel). 2017 Aug 24;9(9):260. doi: 10.3390/toxins9090260. PMID 28837075
- [Background] Park SB, Krishnan AV, Lin CS, Goldstein D, Friedlander M, Kiernan MC. Mechanisms underlying chemotherapy-induced neurotoxicity and the potential for neuroprotective strategies. Curr Med Chem. 2008;15(29):3081-94. doi: 10.2174/092986708786848569. PMID 19075655
- [Background] Rao RD, Michalak JC, Sloan JA, Loprinzi CL, Soori GS, Nikcevich DA, Warner DO, Novotny P, Kutteh LA, Wong GY; North Central Cancer Treatment Group. Efficacy of gabapentin in the management of chemotherapy-induced peripheral neuropathy: a phase 3 randomized, double-blind, placebo-controlled, crossover trial (N00C3). Cancer. 2007 Nov 1;110(9):2110-8. doi: 10.1002/cncr.23008. PMID 17853395
- [Background] Rostami R, Mittal SO, Radmand R, Jabbari B. Incobotulinum Toxin-A Improves Post-Surgical and Post-Radiation Pain in Cancer Patients. Toxins (Basel). 2016 Jan 13;8(1):22. doi: 10.3390/toxins8010022. PMID 26771640
- [Background] Segreto F, Marangi GF, Cerbone V, Persichetti P. The Role of Botulinum Toxin A in the Treatment of Raynaud Phenomenon. Ann Plast Surg. 2016 Sep;77(3):318-23. doi: 10.1097/SAP.0000000000000715. PMID 26808752
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Lavoie Smith EM, Cohen JA, Pett MA, Beck SL. The validity of neuropathy and neuropathic pain measures in patients with cancer receiving taxanes and platinums. Oncol Nurs Forum. 2011 Mar;38(2):133-42. doi: 10.1188/11.ONF.133-142. PMID 21356652
- [Background] Chen WT, Yuan RY, Chiang SC, Sheu JJ, Yu JM, Tseng IJ, Yang SK, Chang HH, Hu CJ. OnabotulinumtoxinA improves tactile and mechanical pain perception in painful diabetic polyneuropathy. Clin J Pain. 2013 Apr;29(4):305-10. doi: 10.1097/AJP.0b013e318255c132. PMID 23462284
- [Background] Ghasemi M, Ansari M, Basiri K, Shaigannejad V. The effects of intradermal botulinum toxin type a injections on pain symptoms of patients with diabetic neuropathy. J Res Med Sci. 2014 Feb;19(2):106-11. PMID 24778662
- [Background] Neumeister MW. Botulinum toxin type A in the treatment of Raynaud's phenomenon. J Hand Surg Am. 2010 Dec;35(12):2085-92. doi: 10.1016/j.jhsa.2010.09.019. PMID 21134617
- [Background] Poole HM, Murphy P, Nurmikko TJ. Development and preliminary validation of the NePIQoL: a quality-of-life measure for neuropathic pain. J Pain Symptom Manage. 2009 Feb;37(2):233-45. doi: 10.1016/j.jpainsymman.2008.01.012. Epub 2008 Aug 3. PMID 18676118
- [Background] Yuan RY, Sheu JJ, Yu JM, Chen WT, Tseng IJ, Chang HH, Hu CJ. Botulinum toxin for diabetic neuropathic pain: a randomized double-blind crossover trial. Neurology. 2009 Apr 28;72(17):1473-8. doi: 10.1212/01.wnl.0000345968.05959.cf. Epub 2009 Feb 25. PMID 19246421
- See also: Botox® [package insert]. Irvine, CA: Allergan, Inc; 2011 — https://www.accessdata.fda.gov/drugsatfda_docs/label/2011/103000s5236lbl.pdf